CLINICAL TRIAL: NCT07235670
Title: Gastrointestinal Hormone Secretion, Bile Acid Homeostasis, Intestinal Permeability and Bacterial Translocation in Primary Biliary Cholangitis (PBC), Primary Sclerosing Cholangitis (PSC), Alcoholic Liver Cirrhosis and Short Bowel Syndrome (SBS)
Brief Title: Gastrointestinal Hormone Secretion, Intestinal Permeability and Short Bowel Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rigshospitalet, Denmark (Other)
Responsible Party: Principal Investigator, Palle Bekker Jeppesen, Principal Investigator, Rigshospitalet, Denmark
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: H-17038155
Record Dates: First submitted 2025-11-14; First posted 2025-11-19 (Actual); Last update posted 2025-11-19 (Actual); Status verified 2025-10

CONDITIONS: Short Bowel Syndrome; Intestinal Resection
Keywords: Gastrin; CCK; GIP; Neurotensin; GLP-1; GLP-2; PYY; Intestinal resection
MeSH Terms: conditions — Short Bowel Syndrome

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Single-arm (Experimental): Standardized meal
  Interventions: Dietary Supplement: Standardized meal

INTERVENTIONS:
Dietary Supplement: Standardized meal — A standardized meal containing 2841 kJ (679 kcal). The meal consisted of 21 g protein, 78 g carbohydrate, and 31 g fat, corresponding to a macronutrient distribution of 13% protein, 46% carbohydrate, and 41% fat. It included 50 g rye bread, 50 g coarse bread, 32 g butter, 40 g cheese (45+), 20 g jam, 150 g fruit yogurt, 100 g banana, and 200 g water

SUMMARY:
The gastrointestinal tract is a complex endocrine organ that regulates a wide range of physiological processes, including those involved in the digestion of nutrients. These processes are dynamically coordinated by specialized cells within the intestinal epithelium which, upon exposure to luminal nutrients, secrete a variety of enteroendocrine hormones, such as Gastrin, Cholecystokinin, Glucose-dependent insulinotropic peptide, Neurotensin, Glucagon-like peptide 1, Glucagon-like peptide 2, and Peptide YY.

In this study, we aim to investigate how resection of different intestinal segments affects fasting and postprandial secretion of these gut hormones, and to characterize how these secretion profiles differ compared with healthy controls.

Patients with a history of intestinal resection will be included and stratified according to the intestinal segments in continuity at the time of study participation into the following anatomical groups:

* Group 1A: Patients with jejunum only in continuity and a total small bowel length <150 cm.
* Group 1B: Patients with an ileostomy and a maximum resection of 30 cm of the terminal ileum. The colon is not in continuity, and the ileocecal valve is also not in continuity.
* Group 2: Patients with <150 cm jejunum anastomosed to the ascending colon or proximally in the transverse colon.
* Group 3: Patients with a jejuno-ileal anastomosis, an intact ileocecal valve, and the entire colon in continuity.

In addition, healthy control subjects will be included to enable comparison between patient groups and normal physiology.

Fasting blood samples will be obtained after a standardized rest period, after which all participants will ingest a standardized meal within 15 minutes. Subsequently, repeated blood samples will be collected at t = 0, 10, 20, 30, 45, 60, 120, 180, and 240 minutes postprandially.

Differences between groups in fasting values, area-under-the-curve (AUC), and incremental AUC, values will be calculated. Differences between anatomical groups will be analyzed using analysis of variance (ANOVA) on log-transformed data to improve model fit. Correlations between the secretion profiles of different enteroendocrine hormones will be assessed using Pearson's r.

ELIGIBILITY:
Inclusion Criteria:

* Having any history of resection of small intestine. Information regarding remnant bowel anatomy will be based on data obtained from patient medical records.
* At least 6 months since last intestinal resection.
* If diagnosed with liver cirrhosis, patients should score a maximum of 12 points on the Child-Pugh scoring system (corresponds to Child-Pugh C with a maximum of 12 points). Patients scoring more than 12 points are considered to have terminal cirrhosis and will be excluded from the study. It is likely that terminally cirrhotic patients have concurrent disease processes that could influence results.
* Age between 18 years and 80 years (both included)
* BMI between 16 and 30 (both included)
* Able to ingest a standardized meal containing 2841 kJ (679 kcal). The meal consisted of 21 g protein, 78 g carbohydrate, and 31 g fat, corresponding to a macronutrient distribution of 13% protein, 46% carbohydrate, and 41% fat. It included 50 g rye bread, 50 g coarse bread, 32 g butter, 40 g cheese (45+), 20 g jam, 150 g fruit yogurt, 100 g banana, and 200 g water

Healthy controls subjects:

* Not diagnosed with any chronic or acute disease
* BMI between 16 and 30 (both included)
* Negative pregnancy test (plasma hCG) for women of childbearing potential (at screening visit)
* Age between 18 years and 80 years (both included)
* Able to ingest the meal presented in inclusion criteria no. 6.

Exclusion Criteria:

* Over hepatic encephalopathy.
* Cholangiocarcinoma.
* Hepatocellular carcinoma.
* Other known or suspected cancer.
* Radiation enteritis, gastrointestinal involvement of systemic scleroderma or other condition of intestinal dysmotility, coeliac disease, refractory or tropical sprue.
* eGFR <30 mL/min/1,73m2
* Clinically meaningful renal disease as judged by the investigator.
* Any condition or disease or circumstance that in the Investigator's opinion would put the patient at any undue risk, prevent completion of the study, or interfere with the analysis of the trial results.
* Positive pregnancy test (plasma hCG) for women of childbearing potential (at screening visit) or lactation.
* Planned to undergo an imminent liver transplantation or have undergone a liver transplantation.
* Positive results on the human immunodeficiency virus (HIV), hepatitis B and/or C tests.
* A history of clinically significant intestinal adhesions and/or chronic abdominal pain.
* History of gallstone within the past 3 years. Gallstones with subsequent cholecystectomy to resolve the issues are acceptable.
* Inflammatory bowel disease (IBD) patients who have NOT been on a stable drug treatment regimen for at least the past 4 weeks.
* Evidence of active IBD in the past 12 weeks.
* Visible blood in the stool within the last 3 months.
* Catheter-related sepsis experienced within the last month.
* Heart failure (New York Heart Association [NYHA] class III-IV) and/or known coronary heart disease defined as unstable angina pectoris and/or myocardial infarction within the last 6 months prior to screening.
* Unplanned hospitalisation of >24 hours duration within 1 month before the screening visit.
* Any use of growth hormone, glutamine or growth factors such as native glucagon-like peptide-2 (GLP-2) or GLP-1 analogues within the last 3 months.
* Any use of dipeptidyl peptidase-4 (DPP-IV) inhibitors within the last 3 months.
* Any use of antibiotics within the last 30 days (except for prophylactic treatment for urinary tract infections).
* Loss of blood or donation of blood or plasma >500 mL within 3 months prior to screening.
* Patient not capable of understanding or not willing to adhere to the trial visit schedules and other protocol requirements.
* For any other reason judged not eligible by the investigator.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2021-06-01 (Actual); Primary Completion 2022-06-16 (Actual); Study Completion 2022-06-16 (Actual)

PRIMARY OUTCOMES:
Fasting and postprandial levels of entero-endocrine hormones | 255 minutes

CONTACTS AND LOCATIONS:
Locations (1):
- Rigshospitalet, Copenhagen, Denmark